CLINICAL TRIAL: NCT03385967
Title: A Randomized, Prospective, Double Blind Clinical Trial to Investigate the Increase in Duration of Analgesia With Addition of 0.25mcg/kg of Dexmedetomidine (DEX) to 25 ml of 0.5%Ropivacaine in Supraclavicular Brachial Plexus Block.
Brief Title: Duration of Analgesia With Dexmedetomidine and Ropivacaine in Brachial Plexus Block
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI is leaving the University of Florida
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201702926
Record Dates: First submitted 2017-12-20; First posted 2017-12-29 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Analgesia; Pain, Acute; Peripheral Nerve Block
Keywords: upper extremity bone fracture
MeSH Terms: conditions — Agnosia; Acute Pain | interventions — Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double blind study of adding dexmedetomidine 0.25mcg/kg body weight to standard dose (25ml) of 0.5%ropivacaine for Brachial plexus block and assessing the analgesia with VAS pain scales (0-10), Satisfaction scale by VAS scale (0-10) and time to first analgesic consumption.
Who Masked: Participant, Care Provider
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ropivacaine only (Active Comparator): 0.5% ropivacaine
  Interventions: Drug: ropivacaine
- ropivacaine with dexmedetomidine (Active Comparator): 25ml of 0.5%ropivacaine with 0.25mcg/kg of dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Drug: ropivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Addition of Dexmedetomidine in block .25mcg/kg of dexmedetomidine
  Other Names: precedex
  Arms: ropivacaine with dexmedetomidine
Drug: ropivacaine — Standard of care 0.5%ropivacaine
  Other Names: naropin

SUMMARY:
This is a prospective, randomized, double blind study of adding dexmedetomidine to ropivacaine for Brachial plexus block and assessing the analgesia with VAS pain scales(0-10), Satisfaction scale by VAS scale(0-10) and time to first analgesic consumption. This study mainly aims to investigate whether addition of dexmedetomidine helps in increasing the duration of analgesia.

DETAILED DESCRIPTION:
In our institute ropivacaine is used for all the peripheral nerve blocks. This a prospective, randomized, double blind clinical trial study comparing the addition of dexmedetomidine vs ropivacaine alone in brachial plexus nerve block. After screening the patient with the inclusion criteria, an informed consent is obtained from the patient by one of the co-investigator.

Adjuvants to local anesthetics are commonly added to prolong the duration of the peripheral nerve block. Sometimes patients have other added comorbidities along with high BMI with history of chronic pain where prolonging the duration of the peripheral nerve block would help with decreased narcotic consumption in the perioperative period with minimal side effects related to the local anesthetics(LA) as well as the adjuncts.

Dexmedetomidine is proven to be better than Clonidine in a recent study. Also perineural dexmedetomidine is proven to be more efficacious compared to intravenous dosing. The investigators are evaluating whether adding dexmedetomidine to standard dose of Ropivacaine helps in prolonging the duration of the peripheral nerve block with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age-18years and above
* Both male and female patients
* BMI->18
* Elective Subacute upper extremity fractures

Exclusion Criteria:

* Chronic pain patients (Pain persisting for more than 3-6months or past the normal healing time of any injury, influences every aspect of a person's quality of life.)
* Patients with drug abuse history in the past 6 months
* ESRD
* Hepatic failure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Duration of Effect | Immediate pre-op until 36hours post block
  To determine the change in duration of analgesia by the time to first intake of analgesic medicine by adding 0.25mcg/kg of dexmedetomidine to 25 ml of 0.5%ropivacaine in Brachial plexus nerve block.

SECONDARY OUTCOMES:
Potential Side Effects | Immediate pre-op until 36hours post block
  To look for the potential side effects of dexmedetomidine like bradycardia and hypotension in the intraoperative and immediate post-operative period.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Ardon, MD, Principal Investigator — University of Florida College of Medicine Jacksonville

IPD SHARING:
Plan to Share IPD: No